CLINICAL TRIAL: NCT06442982
Title: Usefulness of Insole-type Gait Analyzer in Collecting Gait Data From Patients With Gait Disturbance
Brief Title: Analyzing Gait Pattern Using Insole-type Gait Analyzer in Patient With Gait Disturbance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9-2021-0055
Record Dates: First submitted 2024-05-21; First posted 2024-06-05 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Gait Disorders, Neurologic
Keywords: gait analysis; smart insole; neurologic disorder
MeSH Terms: conditions — Gait Disorders, Neurologic; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: This study aims to explore the usefulness of collected data and does not establish a control group. Patients with subjective gait and balance disorders will wear insole-type gait analyzer and walk, then the collected data will be examined."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insole wearing group (Experimental): Patients with subjective gait and balance disorders will wear insole-type gait analyzer and walk, then the collected data will be examined."
  Interventions: Device: insole-type gait analyzer

INTERVENTIONS:
Device: insole-type gait analyzer — Patients with subjective gait and balance disorders will wear insole-type gait analyzer and walk, then the collected data will be examined.

SUMMARY:
The goal of this clinical trial is to explore the usefulness of information from insole-type gait analyzer in adults with subjective gait and balance disorders.

The main questions it aims to answer are:

How useful is an insole-type gait analyzer for collecting gait data from patients with gait disturbances?

Researchers will explore the usefulness of collected data and does not establish a control group.

Participants will:

Participants will conduct survey and perform the Timed up and go test wearing an insole-type gait analyzer.

DETAILED DESCRIPTION:
A screening test is conducted after obtaining consent. The screening test assesses whether participants can walk independently on flat ground, following an inquiry into their baseline symptoms and signs.

Participants will conduct A history survey, a sarcopenia questionnaire, and the International Physical Activity Questionnaire (IPAQ).

Participants will wear insole-type gait analyzer and undergo the Timed Up and Go test.

The measurement values of the accelerometer and pressure sensors recorded in the insole-type gait analyzer will be examined to determine the presence of missing or outlier data. Researchers will explore the data collection frequency and analysis methods to extract clinically significant data.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 19 and over (based on the age on their national ID at the time of consent)
2. adults complaining subjective gait or balance disorders
3. individuals who voluntarily agree to participate in the study and sign a consent form

Exclusion Criteria:

1. individuals unable to walk independently on flat ground for more than 6 minutes
2. individuals who cannot read ordinary print with glasses due to visual reasons
3. individuals who cannot understand conversation even with a hearing aid due to auditory reasons
4. individuals with clinically significant disorders in the cardiovascular, gastrointestinal, respiratory, or endocrine systems
5. individuals considered clinically unsuitable for the trial by the trial manager or person in charge based on significant medical findings.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test (TUG) | TUG test session will last approximately 5 minutes. and TUG test will be performed at baseline.
  The participants will wear insole-type gait analyzer and undergo the Timed Up and Go test.
  The above test assesses walking speed along with balance ability during walking, and this is performed as follows.
  1. A 46 cm high armrest chair, a color cone is placed at a distance of 3 meters from the chair and the subject is instructed to sit on the chair.
  2. In the preparation phase, the subject leans against the chair backrest and places his/her arms on the armrests, then stands up on the instruction "Start", walks 3 meters, turns around the color cone, returns to the starting point and sits down on the chair.
     5) Data Verification The measurement values of the accelerometer and pressure sensors recorded in the insole-type gait analyzer will be examined to determine the presence of missing or outlier data. The investigators will explore the data collection frequency and analysis methods to extract clinically significant data.
Korean version of Sarcopenia Screening Questionnaire | This K-SSQ session will last approximately 1 minutes, it will be performed at baseline.
  Questionnaire that evaluates the decrease in muscle strength and functional performance along with a decrease in muscle mass and it is highly related to aging and chronic diseases. The evaluation method is conducted by having the examiner ask the subject about the following questionnaire, and the scores for the answers are recorded.
  It consists of 5 questions, and each question is scored 0-2 points. The higher the score, the higher the risk of sarcopenia. If the score is 4 or higher, sarcopenia may be suspected.
Korean version of the International Physical Activity Questionnaire (K-IPAQ) | This K-IPAQ session will last approximately 3 minutes, it will be performed at baseline.
  Tests that assess various aspects of an individual's daily physical activity16 and it can provide information about activity level. The examiner questions the subject based on the questionnaire below, records related information, calculates the total activity time and intensity, and classifies it as 'low', 'medium', and 'high'.

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander NB. Differential diagnosis of gait disorders in older adults. Clin Geriatr Med. 1996 Nov;12(4):689-703. PMID 8890111
- [Background] Tinetti ME. Clinical practice. Preventing falls in elderly persons. N Engl J Med. 2003 Jan 2;348(1):42-9. doi: 10.1056/NEJMcp020719. No abstract available. PMID 12510042
- [Background] Bennett DA, Beckett LA, Murray AM, Shannon KM, Goetz CG, Pilgrim DM, Evans DA. Prevalence of parkinsonian signs and associated mortality in a community population of older people. N Engl J Med. 1996 Jan 11;334(2):71-6. doi: 10.1056/NEJM199601113340202. PMID 8531961
- [Background] Salzman B. Gait and balance disorders in older adults. Am Fam Physician. 2010 Jul 1;82(1):61-8. PMID 20590073
- [Background] Verghese J, LeValley A, Hall CB, Katz MJ, Ambrose AF, Lipton RB. Epidemiology of gait disorders in community-residing older adults. J Am Geriatr Soc. 2006 Feb;54(2):255-61. doi: 10.1111/j.1532-5415.2005.00580.x. PMID 16460376
- [Background] Fortin C, Feldman DE, Cheriet F, Labelle H. Clinical methods for quantifying body segment posture: a literature review. Disabil Rehabil. 2011;33(5):367-83. doi: 10.3109/09638288.2010.492066. Epub 2010 Jun 23. PMID 20568973
- [Background] Kim H, Lee S, Lee D, Choi S, Ju J, Myung H. Real-time human pose estimation and gesture recognition from depth images using superpixels and SVM classifier. Sensors (Basel). 2015 May 26;15(6):12410-27. doi: 10.3390/s150612410. PMID 26016921
- [Background] Chun MY. Validity and reliability of korean version of international physical activity questionnaire short form in the elderly. Korean J Fam Med. 2012 May;33(3):144-51. doi: 10.4082/kjfm.2012.33.3.144. Epub 2012 May 24. PMID 22787536

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT06442982/Prot_SAP_001.pdf